CLINICAL TRIAL: NCT04189354
Title: Study of the Synergistic Effects of Biofeedback and Transcranial Electrical Stimulation in Anxio-depressive Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tatiana Besse-Hammer (Other)
Responsible Party: Sponsor-Investigator, Tatiana Besse-Hammer, Head of clinical research unit, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHUB-PSY-COMBINTES 1
Record Dates: First submitted 2019-12-03; First posted 2019-12-06 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Anxiety Depression
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active t-DCS (Experimental): Use of the t-DCS machine with the following stimulation parameters: current intensity of 2mA, electrode size of 25 cm2, duration of stimulation 20 minutes (excluding the fade-in and fade-out periods of 15 seconds).
  Interventions: Device: Transcranial direct current stimulation (t-DCS) device
- Sham t-DCS (Sham Comparator): The condition of use in sham mode follows the same procedure as the active t-DCS except that the active stimulation lasts only 30 seconds at 3mA (60 seconds of active stimulation taking into account the periods of fade in and fade out).
  The stimulator remains switched on during the procedure but does not deliver current. The devices are fully automatic and deliver an active or sham current according to a randomized stimulation code whose meaning is unknown by the operator, in order to respect the triple blind.
  Interventions: Device: Transcranial direct current stimulation (t-DCS) device

INTERVENTIONS:
Device: Transcranial direct current stimulation (t-DCS) device — t-DCS is a brain electrostimulation technique that consists of applying a current of low intensity (between 1 and 2 mA) on the scalp via two electrodes, in order to modify the cerebral activity of the stimulated zones. The investigators use the Soterix Medical t-DCS devices of the mini-CT 1x1 type.

SUMMARY:
Anxio-depressive disorders are characterized by a difficulty in regulating the negative or aversive emotions adequately. These dysfunctions have been linked to a deficit in prefrontal cortex activity. The latter has an inhibitory influence on limbic regions -especially the amygdala- involved in the generation of emotions. By this means, the prefrontal cortex intervenes in the control of the sympathetic and parasympathetic branches of the autonomic nervous system whp are responsible for the physiological components of the emotion, including the variations of the cardiac rhythm (HRV: heart rate variability).

In emotionally demanding situations, the activity of the prefrontal cortex is generally associated with an increase in parasympathetic activity that is exerted by stimulation of the vagus nerve. In patients with anxio-depressive disorder, there is a decrease in the activity of the autonomic nervous system whose variability in heart rate is a recognized marker.

Many studies show a beneficial impact of transcranial direct current stimulation (t-DCS) on anxio-depressive symptoms, particularly when a particular area is targeted: the dorso-lateral prefrontal cortex. The impacts of this intervention are multiple and aim in particular to modulate the activity of the autonomic nervous system to promote regulation.

Biofeedback HRV is a technique that allows you to learn how to modulate your heart rate by means of respiratory control exercises. The patient receives an immediate feedback on the effectiveness of his learning (basic principle of bio-feedback). This intervention will allow to act on the parasympathetic activity and to promote a vagal tone adequate to the emotional regulation. Numerous studies have demonstrated the favorable impact of HRV biofeedback on the reduction of anxious and depressive symptoms.

Since the vagus nerve seems to be a primary pathway in physiologically emotional regulation, and considering that vagal tone can be stimulated by both the activity of the prefrontal cortex and through respiratory control, it appears interesting to study the association of t-DCS with HRV biofeedback techniques.

The first objective of this study is to show that HRV biofeedback training coupled with t-DCS is associated with a greater decrease in anxious symptomatology. The secondary objective of the study is to show that a coupling of these two techniques is associated with an increase of the variability of the cardiac rhythm as well as a more important decrease of the depressive symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of anxio-depressive disorder
* Good understanding of French
* High anxiety level (STAI questionnaire score higher to 46) with reported difficulties to manage this anxiety.

Exclusion Criteria:

* Alcohol dependence (assessed by the AUDIT questionnaire)
* Pregnancy
* t-DCS contra indications : traumatic brain injury, epilepsy, known bipolar disease, electronic or metalic implant
* Known cardiac arrhythmia or intake of beta-blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
State-trait anxiety inventory (STAI-Y) scores | Baseline (day 1)
  Questionnaire with 20 questions, each with 4 possible answers. Each answer corresponds to a score of 1 to 4, 1 indicating the lowest degree of anxiety and 4 the highest degree.
State-trait anxiety inventory (STAI-Y) scores | Day 8
  Questionnaire with 20 questions, each with 4 possible answers. Each answer corresponds to a score of 1 to 4, 1 indicating the lowest degree of anxiety and 4 the highest degree.
State-trait anxiety inventory (STAI-Y) scores | Day 29
  Questionnaire with 20 questions, each with 4 possible answers. Each answer corresponds to a score of 1 to 4, 1 indicating the lowest degree of anxiety and 4 the highest degree.
State-trait anxiety inventory (STAI-Y) scores | One time point between day 60 and day 90
  Questionnaire with 20 questions, each with 4 possible answers. Each answer corresponds to a score of 1 to 4, 1 indicating the lowest degree of anxiety and 4 the highest degree.

SECONDARY OUTCOMES:
Root mean square of successive differences (RMSSD) | Baseline (day 1)
  The Root Mean Square of the Successive Differences (RMSSD) is one of a few time-domain tools used to assess heart rate variability, the successive differences being neighboring RR intervals.
Root mean square of successive differences (RMSSD) | Day 8
  The Root Mean Square of the Successive Differences (RMSSD) is one of a few time-domain tools used to assess heart rate variability, the successive differences being neighboring RR intervals.
Root mean square of successive differences (RMSSD) | Day 29
  The Root Mean Square of the Successive Differences (RMSSD) is one of a few time-domain tools used to assess heart rate variability, the successive differences being neighboring RR intervals.
Root mean square of successive differences (RMSSD) | One time point between day 60 and day 90
  The Root Mean Square of the Successive Differences (RMSSD) is one of a few time-domain tools used to assess heart rate variability, the successive differences being neighboring RR intervals.
High frequency in spectral analysis | Baseline (day 1)
  Spectral analysis of the RR interval is an indirect, noninvasive measurement tool of heart rate variability. High-frequency RR signal (greater than 0.15 Hz) is associated with increased parasympathetic tone, and low-frequency RR signal (0.04-0.15 Hz) is associated with increased sympathetic tone.
High frequency in spectral analysis | Day 8
  Spectral analysis of the RR interval is an indirect, noninvasive measurement tool of heart rate variability. High-frequency RR signal (greater than 0.15 Hz) is associated with increased parasympathetic tone, and low-frequency RR signal (0.04-0.15 Hz) is associated with increased sympathetic tone.
High frequency in spectral analysis | Day 29
  Spectral analysis of the RR interval is an indirect, noninvasive measurement tool of heart rate variability. High-frequency RR signal (greater than 0.15 Hz) is associated with increased parasympathetic tone, and low-frequency RR signal (0.04-0.15 Hz) is associated with increased sympathetic tone.
High frequency in spectral analysis | One time point between day 60 and day 90
  Spectral analysis of the RR interval is an indirect, noninvasive measurement tool of heart rate variability. High-frequency RR signal (greater than 0.15 Hz) is associated with increased parasympathetic tone, and low-frequency RR signal (0.04-0.15 Hz) is associated with increased sympathetic tone.
Montgomery Asberg Depression Rating Scale (MADRS) | Baseline (day 1)
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. A total superior to 20/60 is generally considered abnormal. A level of 30 points is considered a definition of severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) | Day 8
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. A total superior to 20/60 is generally considered abnormal. A level of 30 points is considered a definition of severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) | Day 29
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. A total superior to 20/60 is generally considered abnormal. A level of 30 points is considered a definition of severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) | One time point between day 60 and day 90
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. A total superior to 20/60 is generally considered abnormal. A level of 30 points is considered a definition of severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Cole, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No